CLINICAL TRIAL: NCT06316492
Title: Knowledge, Attitude, and Practice of Viral Hepatitis ( B and C) Among Population in a Village in New Valley Governorate
Brief Title: A Study Done by a Demonstrator and Two Professors in Public Health and Community Medicine Department in Faculty of Medicine in Assiut and New Valley University to Assess Knowledge, Attitude ,and Practice of Rural Population in a Remote Governorate ( New Valley ) Towards Hepatitis B and C Viruses
Acronym: rural_remote
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelrazik Abdellatif Elmewafy, dr, New Valley University
Other Study IDs: 101919039932
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Hepatitis B; Hepatitis C
Keywords: knowledge; attitude; practice; rural; remote; Egypt
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a research aiming to identify knowledge , attitude and practice of population in a village in a remote governorate towards viral hepatitis B and C . It involves home visit interviews with population in this village with the use of questionnaire involving questions asked by the researcher that would be orally answered by the participants to be recorded in papers by the researcher.

DETAILED DESCRIPTION:
PICO : What is the knowledge , practice and attitude of people in a village in a remote governorate towards viral hepatitis B and C ?

Introduction :

There are 5 main strains of the hepatitis virus , named alphabetically A, B, C , D and E and while they share in their ability to cause liver disease , they are different regarding mode of transmission , severity , geographical distribution and methods of prevention (1).

In particular of these 5 strains , both viral hepatitis B and C lead to chronic disease in hundreds of milions of people and are the leading cause of liver cirrhosis , liver cancer and viral hepatitis deaths (2) and good news that a WHO study predicted that four and half million premature viral hepatitis related deaths could be prevented in developing countries by 2030 through vaccination , screening tests , drugs and health education (3 ).

WHO estimated about 300 million people have chronic hepatitis B with chance of about 1.5 new infection yearly (4) with a systematic review and meta analysis of published studies from 2000 to 2022 revealed around 3.67 % prevalence of HBV in overall population in Egypt based on HBsAG with similar incidence in urban and rural areas ,2.4% and 2.15% respectively and the lowest prevalence among children less than 20 years old with history of vaccination aginast HBV as a compulsory vaccination in Egypt thus signifies high vaccination coverage among this age group(5) .

Further steps could be taken to decrease prevalence of HBV in Egypt include blocking chain of infection at mother -infant transmission , increasing the scale of the existing vaccine ,and adopting strategies aiming at screening and treatment(6).

Egypt launched the campaign of "100 Million SIHA" in 2018 and one of the goals of this campaign was screening for viral hepatitis C . After identification of cases through rapid antigen test in this campaign, cases had been directed to further testing and treatment with antiviral medications to cure the infection (6) . The official declaration of progress of Egypt in hepatitis C elimination with reduction in its prevalence10% to 0.38% in overall population in around 10 years has been announced in October 2023 (7) .

Previous study conducted in Egypt in 2013 showed that HCV is more prevalent among lower socioeconomic population sections . The HCV prevalence rate was higher in rural than urban areas with 12% in comparison to 7 % . and in the lowest wealth quintile than the highest quintile with 12% in comparison to 7 % (8). According to another study in 2014 , it showed high transmission rate of HCV in Egypt with each HCV could transmit infection to 3.54 subjects (9).

Although significant improvement in control measures in healthcare settings over the past decade, several areas in the domain of primary prevention have not been adequately addressed , such as limiting HCV transmission via IV drug use , sex workers ,and barbershops and several studies point to a poor knowledge of HCV mode of transmission and management (10) .

Rationale :

There is a need to measure knowledge,attitude , and practice regarding hepatitis virus B and C among population in rural areas of remote governorates as poor knowledge and bad practices are limiting factors in HCV elimination and descreasing HBV prevalance in Egypt

ELIGIBILITY:
Inclusion Criteria:

* Population in a Village in Elkharga in New Valley Governorate aged 18 years and older

Exclusion Criteria:

* 1- Population below age of 18 years 2- Population refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: study will be carried out in a village in Elkharga in New Valley Governorate - the researcher is a demonstrator in Public Health and Community Medicine in faculty of medicine in New Valley University and cons as this village is an example of a village in a remote governorate which is needed to be studied in this research.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess proportion of adequate knowledge , attitude and practice /behaviour towards viral hepatitis B and C in a rural population in New Valley Governorate | 2019-2029
  Using a structured interview questionnaire \El-Ghitany et al.2016 (12) + /El-Ghitany et al Validation of EGCRISC for HCV screening in Egypt (13) as a template measuring :
  1. Sociodemographic characteristics of the studied population
  2. Knowledge of the studied population towards viral hepatitis B and C
  3. Attitude of the studied population towards viral hepatitis B and C
  4. Practice of the studied population towards viral hepatitis B and C through home visits with asked questions to the targeted population by the researcher to be answered orally and then recorded in data entry files by the researcher .

SECONDARY OUTCOMES:
Assess proportion of high risk groups of viral hepatitis B and C in these population thus behaviours made them candidates for viral hepatitis B and C infection | 2019-2029
  Using a structured interview questionnaire \El-Ghitany et al.2016 (12) + /El-Ghitany et al Validation of EGCRISC for HCV screening in Egypt (13) as a template measuring :
  1. Sociodemographic characteristics of the studied population
  2. Knowledge of the studied population towards viral hepatitis B and C
  3. Attitude of the studied population towards viral hepatitis B and C
  4. Practice of the studied population towards viral hepatitis B and C through home visits with asked questions to the targeted population by the researcher to be answered orally and then recorded in data entry files by the researcher .
2- Proportion of health-seeking behaviour of cases ( confirmation of diagnosis, treatment, and follow up ) and proportion of high risk group seeking for screening | 2019-2029
  Using a structured interview questionnaire \El-Ghitany et al.2016 (12) + /El-Ghitany et al Validation of EGCRISC for HCV screening in Egypt (13) as a template measuring :
  1. Sociodemographic characteristics of the studied population
  2. Knowledge of the studied population towards viral hepatitis B and C
  3. Attitude of the studied population towards viral hepatitis B and C
  4. Practice of the studied population towards viral hepatitis B and C through home visits with asked questions to the targeted population by the researcher to be answered orally and then recorded in data entry files by the researcher .

IPD SHARING:
Plan to Share IPD: Undecided
To publish introduction , aim , results , and conclusion of the study after its release

REFERENCES:
- [Background] Azzam A, Khaled H, Elbohy OA, Mohamed SA, Mohamed SMH, Abdelkader AH, Ezzat AA, Elmowafy AOI, El-Emam OA, Awadalla M, Refaey N, Rizk SMA. Seroprevalence of hepatitis B virus surface antigen (HBsAg) in Egypt (2000-2022): a systematic review with meta-analysis. BMC Infect Dis. 2023 Mar 10;23(1):151. doi: 10.1186/s12879-023-08110-5. PMID 36899311
- [Background] Esmat G. Hepatitis C in the Eastern Mediterranean Region. East Mediterr Health J. 2013 Jul;19(7):587-8. No abstract available. PMID 24975301
- [Background] Breban R, Arafa N, Leroy S, Mostafa A, Bakr I, Tondeur L, Abdel-Hamid M, Doss W, Esmat G, Mohamed MK, Fontanet A. Effect of preventive and curative interventions on hepatitis C virus transmission in Egypt (ANRS 1211): a modelling study. Lancet Glob Health. 2014 Sep;2(9):e541-e549. doi: 10.1016/S2214-109X(14)70188-3. Epub 2014 Aug 27. PMID 25304421
- [Background] Hassanin A, Kamel S, Waked I, Fort M. Egypt's Ambitious Strategy to Eliminate Hepatitis C Virus: A Case Study. Glob Health Sci Pract. 2021 Mar 31;9(1):187-200. doi: 10.9745/GHSP-D-20-00234. Print 2021 Mar 31. PMID 33795369
- [Background] El-Ghitany EM, Farghaly AG, Abdel Wahab MM, Farag S, Abd El-Wahab EW. Toward a simple risk assessment screening tool for HCV infection in Egypt. J Med Virol. 2016 Oct;88(10):1767-75. doi: 10.1002/jmv.24520. Epub 2016 Mar 21. PMID 26970264
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] El-Ghitany EM, Farghaly AG, Farag S, Abd El-Wahab EW. Validation of EGCRISC for Chronic Hepatitis C Infection Screening and Risk Assessment in the Egyptian Population. PLoS One. 2016 Dec 21;11(12):e0168649. doi: 10.1371/journal.pone.0168649. eCollection 2016. PMID 28002458
- See also: 1. Omar A. at IOM Egypt , "100 Million SIHA":WHO ,UNHCR and IOM organize screening for Hepatitis C to increase Refugees awareness , IOM (Aug 2019) — https://www.who.int/news/item/09-10-2023-who-commends-egypt-for-its-progress-on-the-path-to-eliminate-hepatitis-c
- See also: 2. WHO editors, Hepatitis, WHO(2023), — https://www.who.int/health-topics/hepatitis
- See also: WHO Eastern Mediterranean Region editors , Egypt becomes the first country to achieve WHO validation on the path to elimination of hepatitis C , WHO Eastern Mediterranean Region (2023), — https://www.emro.who.int/media/news/egypt-becomes-the-first-country-to-achieve-who-validation-on-the-path-to-elimination-of-hepatitis-c.html